CLINICAL TRIAL: NCT07157722
Title: The Potential Role of N-Acetyl Cysteine or Alpha-Lipoic Acid as Adjuvant Therapies in the Treatment of Patients With Beta Thalassemia
Brief Title: Evaluating the Effect of N-Acetyl Cysteine and Alpha Lipoic Acid in Patients With Beta Thalassemia
Acronym: NAC/ALA
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Mahmoud Mohamed Elkholy, Teaching Assistant, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 9250572
Record Dates: First submitted 2025-08-28; First posted 2025-09-05 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Beta Thalassemia
Keywords: NAC; ALA
MeSH Terms: conditions — beta-Thalassemia | interventions — Acetylcysteine; Thioctic Acid

STUDY DESIGN:
Intervention Model Description: This is a randomized, parallel, clinical study that will be conducted on 66 patients with beta-thalassemia who fulfill the selection criteria and will be classified randomly into 3 groups as follows:
  Group I (n = 22):
  This group will include twenty-two patients with beta-thalassemia who will receive conventional thalassemia management (iron chelating agent) only.
  Group II (n = 22):
  This group will include twenty-two patients with beta-thalassemia who will receive conventional thalassemia management (iron chelating agent) plus NAC (600 mg orally once daily) for three months.
  Group III (n = 22):
  This group will include twenty-two patients with beta-thalassemia who will receive conventional thalassemia management (iron chelating agent) plus ALA (600 mg orally once daily) for three months.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group 1: (Iron chelating agent group) (Active Comparator): Patients with beta-thalassemia who will receive conventional thalassemia management (iron chelating agent) only.
  Interventions: Drug: Iron chelating intervention
- Group 2: (Iron chelating agent + NAC group) (Active Comparator): Patients with beta-thalassemia who will receive conventional thalassemia management (iron chelating agent) plus NAC (600 mg orally once daily) for 12 weeks.
  Interventions: Drug: Iron chelating intervention; Drug: N Acetyl cysteine 600mg
- Group 3: (Iron chelating agent + ALA group) (Active Comparator): Patients with beta-thalassemia who will receive conventional thalassemia management (iron chelating agent) plus ALA (600 mg orally once daily) for 12 weeks.
  Interventions: Drug: Iron chelating intervention; Drug: Alpha Lipoic Acid 600 MG Oral Tablets

INTERVENTIONS:
Drug: Iron chelating intervention — JADENU is indicated for the treatment of chronic iron overload due to blood transfusions.
Drug: N Acetyl cysteine 600mg — N-acetyl cysteine (NAC) 600 mg will be administered orally once daily for 12 weeks.
  Arms: Group 2: (Iron chelating agent + NAC group)
Drug: Alpha Lipoic Acid 600 MG Oral Tablets — Alpha lipoic acid (ALA) 600 mg will be administered orally once daily for 12 weeks.
  Arms: Group 3: (Iron chelating agent + ALA group)

SUMMARY:
The current study is to investigate the potential roles of N-acetyl cysteine and Alpha-lipoic acid in patients with beta-thalassemia.

DETAILED DESCRIPTION:
Beta-thalassemia (β-thalassemia) is a hereditary blood disorder, which is characterized by a genetic disorder in the production of β-globin chains. β-thalassemia is inherited mainly by an autosomal recessive manner resulting in reduced synthesis or absence of β-globin chains, leading to ineffective erythropoiesis and chronic hemolytic anemia. It is classified according to the severity into major, intermedia and minor.

This is a randomized, parallel, clinical study that will be conducted on sixty-six patients with beta-thalassemia. The study duration will be 12 weeks. Patients will be divided into three groups as follows:

Group I (n = 22):

This group will include twenty-two patients with beta-thalassemia who will receive conventional thalassemia management (iron chelating agent) only.

Group II (n = 22):

This group will include twenty-two patients with beta-thalassemia who will receive conventional thalassemia management (iron chelating agent) plus NAC (600 mg orally once daily) for three months.

Group III (n = 22):

This group will include twenty-two patients with beta-thalassemia who will receive conventional thalassemia management (iron chelating agent) plus ALA (600 mg orally once daily) for three months.

The study will be approved by the Research Ethical Committee at Faculty of Pharmacy, Tanta University. All participants will be informed about benefits and risks of the study. The privacy of all participants will be respected and the data of enrolled participants will be confidential. All participants will sign their written informed consent.

ELIGIBILITY:
Inclusion Criteria:

* Patients with beta-thalassemia who will receive conventional thalassemia management.
* Both genders.
* Age ≥ 18 years old.

Exclusion Criteria:

* Patients with familial hypercholesterolemia or history of premature atherosclerosis.
* Patients with a prior history of significant cardiovascular diseases, such as coronary artery disease, myocardial infarction, or stroke.
* Patients with severe renal dysfunction.
* Patients with severe hepatic dysfunction.
* Patients with diabetes.
* Patients who will be non-compliant with the prescribed therapy.
* Patients with other hemoglobinopathies.
* Pregnant women.
* Obese patients.
* Patients who will receive antioxidant or anti-inflammatory medications.
* Patients with inflammatory diseases, such as Systemic lupus erythematous, rheumatoid arthritis and inflammatory bowel disease.
* Patients with oxidative stress related diseases, such as Alzheimer, Parkinson, COPD and cancer.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2025-08-30 (Estimated); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
The change from baseline in carotid intima media thickness (CIMT) | 3 months
  Non-invasive imaging technique, such as carotid ultrasonography will be used to measure carotid intima media thickness

SECONDARY OUTCOMES:
Change in Malondialdehyde (MDA) | 3 months
  Malondialdehyde (MDA) level will be assessed using commercially available kit
Change in high sensitivity C-reactive protein (hs-CRP) | 3 months
  High sensitivity C-reactive protein (hs-CRP) level will be assessed using commercially available kit.
Change in asymmetric dimethyl arginine (ADMA) | 3 months
  Asymmetric dimethyl arginine (ADMA) level will be assessed using commercially available kit.
Change in lipid profile | 3 months
  HDL, total cholesterol and triglycerides will be assessed using commercially available kits.

CONTACTS AND LOCATIONS:
Overall Officials: Sahar M El-Haggar, Professor, Study Director — Tanta University; Tarek M Mostafa, Professor, Study Director — Tanta University; Basma A Mansour, Lecturer, Study Director — Faculty of Medicine - Mansoura University; Mohammed A El hawary, Assistant Professor, Principal Investigator — Faculty of Medicine - Mansoura University; Mahmoud M Elkholy, Teaching Assistant, Principal Investigator — Tanta University
Locations (1):
- Faculty of Pharmacy - Tanta University, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: No